CLINICAL TRIAL: NCT02331277
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Subcutaneous Doses of BI 655064 in Healthy Chinese Male Volunteers (Randomised, Double-blind, Placebo-controlled, Clinical Phase I Study)
Brief Title: Safety and Pharmacokinetics of Multiple Doses of BI 655064 in Healthy Chinese Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1293.9
Record Dates: First submitted 2015-01-05; First posted 2015-01-06 (Estimated); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-09

CONDITIONS: Healthy
MeSH Terms: interventions — BI 655064

ARMS (2):
- BI 655064 (Experimental): Subjects received BI 655064 240 milligram (mg) via subcutaneous injection every week, until 4 weeks.
  Interventions: Drug: BI 655064
- Placebo (Placebo Comparator): Subjects received placebo matching to BI 655064 via subcutaneous injection every week, until 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 655064 — subcutaneous injection
  Arms: BI 655064
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of multiple doses of BI 655064 following weekly subcutaneous injection for 4 weeks in healthy Chinese male volunteers.

The secondary objective is the exploratory evaluation of the pharmacokinetics and pharmacodynamics of multiple doses of BI 655064 following weekly subcutaneous injection for 4 weeks in healthy Chinese male volunteers.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males according to the investigator's assessment, as based on the following criteria: a complete medical history including a physical examination, vital signs (Blood pressure, Pulse rate), 12-lead Echocardiogram, and clinical laboratory tests
2. Chinese ethnicity according to the following criteria:

   Ethnic Chinese, born in China or ethnic Chinese born outside of China, and a descendent of 4 ethnic Chinese grandparents who were all born in China
3. Age within the range of 20 to 45 years inclusive
4. Body Mass Index within the range of 18.5 and 25 kg/m2 inclusive
5. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation
6. Male subjects who

   * are documented to be sterile or consistently and correctly use a condom while their female partners (if of childbearing potential) agree to use any of the following adequate contraception methods: implants, injectables, combined oral contraceptives, intrauterine device (IUD) from the date of screening until at least 6 months after the last dose of BI 655064 taken in the current trial.
   * do not donate any sperm sample for procreation purposes, from the date of screening until at least 6 months after last dose of BI 655064 taken in the current trial.

It is the responsibility of the male subject to ensure that his partner does not become pregnant during all the study duration.

Exclusion criteria:

1. Any finding in the medical examination (including Blood pressure, Pulse rate or Echocardiogram) deviating from normal and judged clinically relevant by the investigator
2. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
3. Any evidence of a concomitant disease judged clinically relevant by the investigator
4. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
5. Diseases of the central nervous system (such as epilepsy), other neurological disorders or psychiatric disorders
6. History of relevant orthostatic hypotension, fainting spells, or blackouts
7. History of relevant allergy/hypersensitivity (including allergy to the trial medication or its excipients)
8. Intake of drugs with a long half-life (>24 hours) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication
9. Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial
10. Participation in another trial with investigational drug administration within 60 days prior to administration of trial medication
11. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes/day)
12. Inability to refrain from smoking on trial days
13. Alcohol abuse (consumption of more than 20 g/day)
14. Drug abuse or positive drug screen
15. Blood donation (more than 100 mL within 30 days prior to administration of trial medication or intended during the trial)
16. Intention to commence new exercise regimen or excessive physical activities within one week prior to administration of trial medication or during the trial
17. Inability to comply with protocol requirements (including dietary regimen of trial site) as assessed by the investigator
18. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of QTc interval > 450 ms) at screening examination
19. Positive results of infectious serology (Hepatitis B Surface Antigen, Hepatitis B Core Antibody, Hepatitis C Antibody or Human Immunodeficiency Virus) at screening examination
20. History of tuberculosis infection and/or positive Quantiferon Tuberculosis-Gold test at screening examination
21. Abnormal results of coagulation values indicating an increased risk for bleeding or thromboembolism or complicating the safety evaluation during the study as determined by the investigator at screening examination
22. Subjects who in the investigator's judgement are perceived as having an excessive risk of thromboembolism for example because of a personal history and/or a first degree relative with a personal history with onset under the age of 55 of significant thromboembolism, including but not limited to deep vein thrombosis, pulmonary embolism, cortical sinus thrombosis, coronary and cerebrovascular events, and peripheral arterial insufficiency.
23. Deficiency of antithrombin III or protein S or protein C at screening examination
24. Prolongation of bleeding time out of reference range at screening examination
25. Subject is assessed by the investigator as unsuitable for inclusion e.g. considered not able to understand and comply with study requirements or has a condition that would not allow safe participation in the study

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-05-25 (Actual); Study Completion 2016-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1293.9.8201 Boehringer Ingelheim Investigational Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, double-blind, placebo-controlled, multiple dose trial.
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the clinical trial at any time for any reason given. Close monitoring of all subjects was adhered to throughout the trial conduct. Rescue medication was allowed for all patients as required.
Period: Overall Study
Arm/Group | Placebo | BI 655064
Started | 3 | 9
Completed | 2 | 9
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This set included all subjects who were dispensed study medication and were documented to have received at least 1 dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 655064 | Total
Number analyzed (Participants) | 3 | 9 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.0 (4.36) | 25.1 (3.41) | 26.1 (3.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 9 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 9 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 9 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug-related Adverse Events.
Description: Percentage of subjects with drug-related adverse events (AEs). Medical judgment was used to determine the relationship between study medication and AEs, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.
Time Frame: From the first drug administration until 126 days after last drug administration, up to 148 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of subjects
Arm/Group | Placebo | BI 655064
Number analyzed (Participants) | 3 | 9
Percentage of subjects | 66.7 | 55.6

2. Secondary Outcome: Maximum Measured Concentration of BI 655064 in Plasma After the 1st Dose (Cmax)
Description: Maximum measured concentration of BI 655064 in plasma after the 1st dose (Cmax).
Time Frame: Pharmacokinetic samples were collected at -3, 8, 12, 24, 48, 72, 84, 96, 108, 120, 144 and 167.5 hours (h) after first drug administration on day 1.
Population: The pharmacokinetic (PK) set (PKS): This set included all evaluable subjects in TS who provided at least 1 PK parameter. One subject was excluded from the PKS as he developed a positive anti-BI 655064 antibodies response.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram (μg) / milliLitre (mL)
Arm/Group | BI 655064
Number analyzed (Participants) | 8
microgram (μg) / milliLitre (mL) | 22.9 (72.3)

3. Secondary Outcome: Time From Dosing to Maximum Measured Concentration of BI 655064 in Plasma After the 1st Dose (Tmax)
Description: Time from dosing to maximum measured concentration of BI 655064 in plasma after the 1st dose (tmax).
Time Frame: Pharmacokinetic samples were collected at -3, 8, 12, 24, 48, 72, 84, 96, 108, 120, 144 and 167.5 h after first drug administration on day 1.
Population: PKS. One subject was excluded from the PKS as he developed a positive anti-BI 655064 antibodies response.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | BI 655064
Number analyzed (Participants) | 8
hours (h) | 132 [72 to 168]

4. Secondary Outcome: Area Under the Concentration-time Curve of BI 655064 in Plasma After the 1st Dose Over a Uniform Dosing Interval τ (AUCτ,1)
Description: Area under the concentration-time curve of BI 655064 in plasma after the 1st dose over a uniform dosing interval τ (= 1 week) (AUCτ,1).
Time Frame: as for outcome 3
Population: PKS. One subject was excluded from the PKS as he developed a positive anti-BI 655064 antibodies response.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | BI 655064
Number analyzed (Participants) | 8
μg*h/mL | 2610 (79)

5. Secondary Outcome: Maximum Measured Concentration of BI 655064 in Plasma After the 4th Dose (Cmax,4)
Description: Maximum measured concentration of BI 655064 in plasma after the 4th dose (Cmax,4).
Time Frame: Pharmacokinetic samples were collected at 505, 516, 528, 552, 576, 600, 624, 648, 672, 696, 744, 816, 912, 1008, 1176, 1344, 1512, 1848, 2520 and 3192 h after fourth drug administration on day 22.
Population: PKS. One subject was excluded from the PKS as he developed a positive anti-BI 655064 antibodies response.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | BI 655064
Number analyzed (Participants) | 8
μg/mL | 74.1 (50.4)

6. Secondary Outcome: Time From Dosing to Maximum Measured Concentration of BI 655064 in Plasma After the 4th Dose (Tmax,4)
Description: Time from dosing to maximum measured concentration of BI 655064 in plasma after the 4th dose (tmax,4).
Time Frame: as for outcome 5
Population: PKS. One subject was excluded from the PKS as he developed a positive anti-BI 655064 antibodies response.
Measure: Median (Full Range); unit: h
Arm/Group | BI 655064
Number analyzed (Participants) | 8
h | 84.2 [12 to 144]

7. Secondary Outcome: Area Under the Concentration-time Curve of BI 655064 in Plasma After the 4th Dose Over a Uniform Dosing Interval τ (AUCτ,4)
Description: Area under the concentration-time curve of BI 655064 in plasma after the 4th dose over a uniform dosing interval τ (= 1 week) (AUCτ,4).
Time Frame: as for outcome 5
Population: PKS. One subject was excluded from the PKS as he developed a positive anti-BI 655064 antibodies response.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | BI 655064
Number analyzed (Participants) | 8
μg*h/mL | 10900 (49.9)

8. Secondary Outcome: Accumulation Ratio of BI 655064 in Plasma After Administration of the 4th Dose Over the Dosing Interval τ, Expressed as Ratio of Cmax After the 4th Dose and After the 1st Dose (RA,Cmax,4)
Description: Accumulation ratio of BI 655064 in plasma after administration of the 4th dose over the dosing interval τ (= 1 week), expressed as ratio of Cmax after the 4th dose and after the 1st dose (RA,Cmax,4).
Time Frame: Pharmacokinetic samples were collected at -3, 8, 12, 24, 48, 72, 84, 96, 108, 120, 144 and 167.5 h for Cmax and 505, 516, 528, 552, 576, 600, 624, 648, 672, 696, 744, 816, 912, 1008, 1176, 1344, 1512, 1848, 2520, 3192 and 5880 h for Cmax,4.
Population: PKS. One subject was excluded from the PKS as he developed a positive anti-BI 655064 antibodies response.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Cmax after the 4th and 1st dose
Arm/Group | BI 655064
Number analyzed (Participants) | 8
Ratio of Cmax after the 4th and 1st dose | 3.24 (24.8)

9. Secondary Outcome: Accumulation Ratio of BI 655064 in Plasma After Administration of the 4th Dose Over the Dosing Interval τ, Expressed as Ratio of AUC After the 4th Dose and After the 1st Dose (RA,AUC,4)
Description: Accumulation ratio of BI 655064 in plasma after administration of the 4th dose over the dosing interval τ (= 1 week), expressed as ratio of AUC after the 4th dose and after the 1st dose (RA,AUC,4).
Time Frame: Pharmacokinetic samples were collected at -3, 8, 12, 24, 48, 72, 84, 96, 108, 120, 144 and 167.5 h for AUCτ,1 and 505, 516, 528, 552, 576, 600, 624, 648, 672, 696, 744, 816, 912, 1008, 1176, 1344, 1512, 1848, 2520, 3192 and 5880 h for AUCτ,4.
Population: PKS. One subject was excluded from the PKS as he developed a positive anti-BI 655064 antibodies response.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC after the 4th and 1st dose
Arm/Group | BI 655064
Number analyzed (Participants) | 8
Ratio of AUC after the 4th and 1st dose | 4.19 (32.9)

ADVERSE EVENTS:
Time Frame: From the first drug administration until 126 days after last drug administration, up to 148 days.
Arm/Group | Placebo | BI 655064
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/9
Other Adverse Events (participants affected / at risk) | 3/3 | 6/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | BI 655064 (N=9)
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Breath odour (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 2
Fatigue (General disorders) | 0 | 1
Injection site bruising (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0
Affect lability (Psychiatric disorders) | 1 | 0
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.